CLINICAL TRIAL: NCT02126241
Title: The Use of Impedance-Based Non-invasive Cardiac Output Measurement (NICaS) for Optimizing Cardiac Resynchronization Therapy: a Pilot Clinical Trial.
Brief Title: Non-Invasive Cardiac Output Measurement for CRT Optimization
Acronym: NICaS-CRT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sheba Medical Center (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SHEBA-1176-14-MG-CTIL
Record Dates: First submitted 2014-04-27; First posted 2014-04-29 (Estimated); Last update posted 2015-08-06 (Estimated); Status verified 2015-08

CONDITIONS: Congestive Heart Failure
Keywords: Heart Failure; Cardiac Resyncronization Therapy; Optimization; Non-invasive cardiac system; Impedance measured cardiac output
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- NICaS guided CRT optimization (Experimental): For each subject, we will determine a set of AV and VV delays values, for which the NICaS measured CO will be maximum. In each patient, the CRT device will then be programmed according to these values.
  Interventions: Other: NICaS guided CRT optimization

INTERVENTIONS:
Other: NICaS guided CRT optimization — 1. Baseline CO measurement by NICaS
  2. AV delay optimization:
     1. AV delay will be changed (increase and decrease) by 30 ms steps , and for each new AV value, the CO will be real-time measured by NICaS
     2. The AV delay yielding the maximal CO, will be considered the optimal AV delay
     3. The device will be programmed using the optimal AV delay
  3. VV delay optimization:
     1. After Step 2, the baseline VV delay will be changed (increase and decrease; meaning that we will be pacing alternatively the LV before the RV, then the RV before the LV), by 30 ms steps, and for each new VV value, the CO will be real-time measured by NICaS
     2. The VV delay yielding the maximal CO, will be considered the optimal VV delay
     3. The device will be programmed using the optimal VV delay

SUMMARY:
This proposal aims to evaluate the added clinical and echocardiographic benefit of using the non-invasive impedance-based cardiac output measurement system (NICaS) for optimizing atrio-ventricular and inter-ventricular delays in chronic (more than 6 months) CRT recipients.

DETAILED DESCRIPTION:
1. Introduction

   Cardiac resynchronization therapy (CRT) is an efficient treatment in heart failure (HF) patients with left ventricular (LV) systolic dysfunction and wide QRS. It is associated with improved exercise capacity, quality of life and left ventricular ejection fraction, as well as reverse remodeling, mitral regurgitation reduction, and mortality reduction.

   Predicting response to CRT is important as 30% of patients have no or minimal clinical improvement following CRT. Several parameters have been shown to influence response following implantation. Some relate to patients' characteristics including underlying heart disease, comorbidities and arrhythmias, type and severity of conduction disorder, presence and degree of dyssynchrony, presence and extent of scar tissue and functional myocardial reserve. Others are associated with technical aspects, including electrical and anatomical positioning of LV lead, programming mode and percentage of effective bi-ventricular pacing.

   Optimization of the atrio-ventricular (AV) delay and inter-ventricular (VV) delays can be used for maximizing CRT benefit, but is not routinely recommended by current guidelines. Standard optimization is performed under echocardiography guidance - a time and resource consuming method. Other non-invasive methods, such as impedance cardiography, can be used for AV delay optimization.
2. Rationale for CRT optimization using NICaS

   The non-invasive cardiac system (NICaS) is a whole-body bioimpedance measurement method allowing real-time cardiac output (CO) assessment. It has been FDA approved for assisting in the diagnosis, monitoring and care management of patients with congestive heart failure as well as for cardiac pacemaker optimization. Clinical trials have shown its utility for the follow-up of outpatient monitoring chronic heart failure, for monitoring patients with heart failure and pulmonary hypertension.

   NICaS is sensitive enough for detecting real-time small changes in CO. Based on NICaS measured CO changes following AV and VV delays modifications, small series support its use for CRT optimization in a clinical setting, suggesting it may be associated with a reduction in non-responder rate.
3. Hypothesis

   We hypothesize that the use of NICaS for optimization of AV and VV delays in chronic (more than 6 months) CRT recipients may result in an added clinical and echocardiographic benefit.
4. Specific Aims

   1. Identify the CRT recipients who are prone to benefit following CRT optimization, by finding the predictors (clinical, ECG, echocardiographic, hemodynamic) for significant cardiac output improvement after NICaS guided CRT optimization
   2. Correlate the degree of cardiac output improvement (as measured by NICaS) after NICaS guided CRT optimization, with clinical and echocardiographic changes at 6 months
5. Timeline:

I. At Inclusion

I.A. Baseline assessment. Patients included in the study will benefit from the following at baseline assessment, performed in an outpatient setting:

1. Clinical evaluation:

   1. history;
   2. NYHA class; six-minute walk test (6MWT); Minnesota Living with Heart Failure questionnaire for the quality of life (QoL);
   3. status following CRT (responder/non-responder);
   4. physical evaluation;
   5. current medication
2. ECG
3. Device interrogation
4. Transthoracic echocardiography (including dyssynchrony parameters)

I.B. NICaS protocol for optimal AV and VV delays assessment. After baseline assessment is completed, patients will benefit from NICaS hemodynamic assessment and CRT programming according to NICaS guided optimal AV and VV delays. (for NICaS protocol for optimal AV and VV delays measurements - see Interventions)

I.C. After NICaS guided CRT programming, patients will perform a 6MWT

II. At 6 months follow-up. At 6 months, patients will benefit from the following evaluations:

1. Clinical: NYHA class, 6MWT, Minnesota Living with Heart Failure questionnaire for the quality of life, current medication
2. ECG
3. Device interrogation
4. Transthoracic echocardiography

ELIGIBILITY:
Inclusion Criteria:

* Patients implanted with a CRT device at least 6 months before, in concordance with AHA/ACC or ESC/EHRA Guidelines (Class I or II) for CRT implantation
* NYHA class I - III heart failure
* Stable sinus rhythm
* Bi-ventricular pacing ≥ 90%
* Patient provides informed consent.

Exclusion Criteria:

* NYHA class IV heart failure
* Permanent or persistent atrial fibrillation
* Bi-ventricular pacing <90%
* Inability to perform the six-minute walk test

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2014-04; Primary Completion 2014-11 (Actual); Study Completion 2015-05 (Actual)

PRIMARY OUTCOMES:
Predictors for significant cardiac output improvement | Within the first year after beginning of study
  Using logistic regression, we will look for predictors (clinical, ECG, echocardiographic, hemodynamic) of significant (at least 20%) acute cardiac output improvement (as assessed by NICaS), after NICaS guided AV and VV delays optimization.

SECONDARY OUTCOMES:
Acute six-minute walk test changes after NICaS optimization | Within the first 24 hours after enrollment
  After NICaS guided AV and VV delays optimization, each patient will perform a six-minute walk test, which will be compared to the baseline (before NICaS optimization) six-minute walk test. A 10% change will be considered significant.
Reverse remodeling | At 6 months after enrollment
  Each patient will undergo routinely a 6-month echocardiography which will be compared to the baseline (inclusion day) echocardiography. A relative reduction of 10% of the left ventricular end-systolic volume will be considered as positive reverse remodeling.
Hospitalization rate for heart failure | Within the first 6 months after enrollment
  Hospitalization rate for acute heart failure during the first 6 months following NICaS guided CRT optimization
Supraventricular arrhythmia occurrence | At 6 months after enrollment
  CRT device measurement of the total time spent in auto-mode switch during the first 6 months following NICaS guided CRT optimization, and comparison to the 6 months prior to the optimization.
Clinical improvement | At 6 months after enrollment
  Clinical improvement at 6 months after CRT optimization will be assessed using a composite score combining NYHA class, QoL and the 6MWT.
  Each will be classified as improved (+1), stable (0) or worsened (-1) and the three components will be summed. The patient will be considered improved if he will have had ≥1 class reduction in his NYHA class, worsened if he will have had ≥1 class increase and unchanged if he will have had no change in his baseline NYHA class. Similar definitions will be used for absolute variation (improvement or deterioration) of 10 points in QoL, or relative 10%change in six-minute walk distance.
  A clinical improvement will be considered in the presence of a summed score ≥+1 without death during the first 6 months of follow-up after CRT optimization.

CONTACTS AND LOCATIONS:
Overall Officials: Michael Glikson, MD, Principal Investigator — Sheba Medical Center
Locations (1):
- Sheba Medical Center, Ramat Gan, Israel

REFERENCES:
- [Background] Brignole M, Auricchio A, Baron-Esquivias G, Bordachar P, Boriani G, Breithardt OA, Cleland J, Deharo JC, Delgado V, Elliott PM, Gorenek B, Israel CW, Leclercq C, Linde C, Mont L, Padeletti L, Sutton R, Vardas PE; ESC Committee for Practice Guidelines (CPG); Zamorano JL, Achenbach S, Baumgartner H, Bax JJ, Bueno H, Dean V, Deaton C, Erol C, Fagard R, Ferrari R, Hasdai D, Hoes AW, Kirchhof P, Knuuti J, Kolh P, Lancellotti P, Linhart A, Nihoyannopoulos P, Piepoli MF, Ponikowski P, Sirnes PA, Tamargo JL, Tendera M, Torbicki A, Wijns W, Windecker S; Document Reviewers; Kirchhof P, Blomstrom-Lundqvist C, Badano LP, Aliyev F, Bansch D, Baumgartner H, Bsata W, Buser P, Charron P, Daubert JC, Dobreanu D, Faerestrand S, Hasdai D, Hoes AW, Le Heuzey JY, Mavrakis H, McDonagh T, Merino JL, Nawar MM, Nielsen JC, Pieske B, Poposka L, Ruschitzka F, Tendera M, Van Gelder IC, Wilson CM. 2013 ESC Guidelines on cardiac pacing and cardiac resynchronization therapy: the Task Force on cardiac pacing and resynchronization therapy of the European Society of Cardiology (ESC). Developed in collaboration with the European Heart Rhythm Association (EHRA). Eur Heart J. 2013 Aug;34(29):2281-329. doi: 10.1093/eurheartj/eht150. Epub 2013 Jun 24. No abstract available. PMID 23801822
- [Background] Delnoy PP, Ritter P, Naegele H, Orazi S, Szwed H, Zupan I, Goscinska-Bis K, Anselme F, Martino M, Padeletti L. Association between frequent cardiac resynchronization therapy optimization and long-term clinical response: a post hoc analysis of the Clinical Evaluation on Advanced Resynchronization (CLEAR) pilot study. Europace. 2013 Aug;15(8):1174-81. doi: 10.1093/europace/eut034. Epub 2013 Mar 14. PMID 23493410
- [Background] Tanino Y, Shite J, Paredes OL, Shinke T, Ogasawara D, Sawada T, Kawamori H, Miyoshi N, Kato H, Yoshino N, Hirata K. Whole body bioimpedance monitoring for outpatient chronic heart failure follow up. Circ J. 2009 Jun;73(6):1074-9. doi: 10.1253/circj.cj-08-0847. Epub 2009 Apr 16. PMID 19372625
- [Background] Heinroth KM, Elster M, Nuding S, Schlegel F, Christoph A, Carter J, Buerke M, Werdan K. Impedance cardiography: a useful and reliable tool in optimization of cardiac resynchronization devices. Europace. 2007 Sep;9(9):744-50. doi: 10.1093/europace/eum086. Epub 2007 May 11. PMID 17496288
- [Background] Turcott RG, Witteles RM, Wang PJ, Vagelos RH, Fowler MB, Ashley EA. Measurement precision in the optimization of cardiac resynchronization therapy. Circ Heart Fail. 2010 May;3(3):395-404. doi: 10.1161/CIRCHEARTFAILURE.109.900076. Epub 2010 Feb 22. PMID 20176716